CLINICAL TRIAL: NCT05209750
Title: Pilot Study of FAPI PET/CT for Locoregional (re)Staging of Lymph Nodes in Colorectal Carcinoma
Brief Title: FAPI PET/CT for Lymph Node Staging in Colorectal Carcinoma
Acronym: FAPI-CRC1
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Netherlands Cancer Institute (Other)
Collaborators: Noordwest Ziekenhuisgroep (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: M21PFP
Record Dates: First submitted 2022-01-13; First posted 2022-01-27 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: Colorectal Cancer
Keywords: Lymph node; Staging; FAPI; PET/CT; Rectal cancer; Colon cancer
MeSH Terms: conditions — Colorectal Neoplasms; Rectal Neoplasms; Colonic Neoplasms

STUDY DESIGN:
Intervention Model Description: Interventional study without concurrent controls
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- FAPI PET/CT (Experimental): Colon cancer patients: one FAPI PET/CT scan early after standard diagnostic imaging and prior to planned surgery.
  Rectal cancer patients: two FAPI PET/CT scans, one for initial staging (pre neoadjuvant therapy) and one for restaging (post neoadjuvant therapy).
  Interventions: Diagnostic Test: FAPI PET/CT

INTERVENTIONS:
Diagnostic Test: FAPI PET/CT — This study applies the radiopharmaceutical 18Fluor-FAPI-74 (shortly called FAPI) for molecular imaging of FAP expression in vivo with FAPI PET/CT, to assess the presence and distribution of activated tumour-associated fibroblasts as a marker of tumour stroma and indirectly as a marker of CRC.
  Other Names: Fluor-18-FAPI-74

SUMMARY:
To describe the accuracy of FAPI PET/CT in the detection of regional lymph node metastases in patients with colorectal cancer in comparison with standard diagnostic imaging and (in operated patients) histopathology, aiming to provide early evidence of the diagnostic value of FAPI PET/CT.

DETAILED DESCRIPTION:
Rationale: In patients with colorectal cancer the detection of small nodal metastases with standard diagnostic imaging (CT and/or MRI) is challenging. This may result in suboptimal staging and ultimately in suboptimal treatment. Colorectal cancer is typically associated with a tumour stroma containing large numbers of activated tumour-associated fibroblasts. Radiolabelled fibroblast activation protein inhibitor (FAPI) compounds bind selectively to these fibroblasts, and thereby allow sensitive and specific imaging of tumour stroma with FAPI PET/CT. Recently published research has indicated that FAPI PET/CT can accurately detect macroscopic colorectal cancer lesions. We have recently demonstrated that tumour stroma also develops in lymph node metastases with a tumour diameter of just a millimetre. Improved detection in the primary tumour area and in regional lymph nodes provided by FAPI PET/CT may contribute to more accurate staging with potential impact on patient management e.g., selection for neoadjuvant treatment. However, until now FAPI PET/CT has mainly been used to visualise tumour in metastatic patients with various tumour types in the scope of palliative treatment, and its specific diagnostic value for detection and locoregional staging of colorectal cancer is currently unknown. We will now use FAPI PET/CT in a pilot study to explore the potential diagnostic value in the detection of regional lymph node metastases, and to identify opportunities for further prospective research in the areas of diagnostics, radiotherapy, and FAPI-based theragnostic therapy.

Objective: To describe the accuracy of FAPI PET/CT in the detection of regional lymph node metastases in patients with colorectal cancer in comparison with standard diagnostic imaging and (in operated patients) histopathology, aiming to provide early evidence of the diagnostic value of FAPI PET/CT.

Study design: Multicentre prospective cross-sectional diagnostic pilot study. Study population: The study involves 30 patients with newly detected clinically node positive colorectal cancer stratified by 20 patients with colon cancer and 10 patients with rectal cancer. All patients undergo local treatment of the primary colorectal tumour.

Intervention: Participants receive standard diagnostic imaging with contrast enhanced CT thorax-abdomen (all patients) and pelvic MRI for initial staging and restaging after neoadjuvant treatment (rectal cancer patients only). In patients with colon cancer, one FAPI PET/CT scan is added as a diagnostic intervention in the scope of this study early after standard diagnostic imaging and prior to planned surgery. In patients with rectal cancer, two FAPI PET/CT scans are added as diagnostic interventions i.e., for initial staging and restaging (pre and post neoadjuvant therapy). The FAPI PET/CT results will not guide treatment decisions.

Main study parameters: The main objective is to describe the diagnostic accuracy of FAPI PET/CT in detecting regional lymph node metastases relative to standard of care diagnostic imaging. FAPI PET/CT will be visually correlated with contrast-enhanced CT in colon cancer patients, and pelvic MRI pre- and post-neoadjuvant treatment in rectal cancer patients. Histopathology of the resected specimen will serve as reference test for operated patients. Secondary outcomes include description of additional findings on FAPI PET/CT, correlation between tumour stroma in resected lymph node metastases and tracer uptake of regional lymph nodes on FAPI PET/CT, and evaluation of response to neoadjuvant treatment on FAPI PET/CT in rectal cancer. All outcomes are descriptive and serve as pilot for a potential subsequent larger prospective diagnostic study.

Nature and extent of the burden and risks associated with participation, benefit, and group relatedness: Participation in this study has no significant risks and will not induce a delay in diagnosis or treatment because the outcomes of the FAPI PET/CT will not guide treatment decisions. The FAPI PET/CT scan involves a total procedure duration of maximally 2 hours and an estimated radiation dose of 6 mSv per procedure (3 mSv for an administered dose of 200 MBq Fluor-18-FAPI, and 3 mSv for the associated low dose CT scan). This radiation dose (6 mSv in colon cancer patients of > 18 years and 12 mSv in rectal cancer patients of > 50 years) is well within the range of normal diagnostic procedures and does not induce a significant risk in the selected population with colorectal cancer. In addition, the Fluor-18-FAPI radiopharmaceutical is thus far not associated with side effects after injection.

ELIGIBILITY:
Inclusion Criteria:

* Biopsy proven newly detected adenocarcinoma of the colon or rectum
* cTany N1-2 Many using TNM 8th edition and based on standard diagnostic imaging including contrast enhanced-CT thorax-abdomen (for colon and rectum) and pelvic MRI (for rectum)
* Indication for curative local treatment of the primary colon/rectal tumour
* Signed written informed consent prior to any study specific procedure

For colon cancer patients:

* Age > 18 years
* Indication for surgery including resection of the colon tumour and the corresponding mesentery
* Surgery can be planned within 5 weeks after diagnostic imaging
* Surgery takes place in one of the participating centres of this study

For rectal cancer patients:

* Age > 50 years and older
* Indication for neoadjuvant (chemo)radiotherapy of the rectal tumour
* Planned for response assessment after (chemo)radiotherapy with pelvic MRI
* Planned for surgery or an organ preservation approach in one of the participating centres of this study * Related to the allowed radiation dose per age category for diagnostic imaging and in accordance with the guideline of the Dutch Commission for Radiation Dosimetry (NCS).

Exclusion Criteria:

* Inability to provide informed consent
* Histopathology of mucinous adenocarcinoma
* WHO > 2
* Pregnancy
* Lactation, unable to substitute for 24 hours after FAPI PET/CT
* Known second malignant disease that may complicate image interpretation including a second primary at time of colorectal cancer diagnosis
* Inability to cooperate with the scan process: inability to lie relatively still and in supine for 30-60 minutes or patient body habitus above scanner dimensions
* Suspicion of peritoneal metastases based on contrast-enhanced CT and/or MRI
* Treatment setting without local treatment of the primary colorectal tumour

For colon cancer patients:

* Absence of diagnostic contrast enhanced-CT thorax-abdomen
* Refusal of surgery by the patient
* Indication for neoadjuvant treatment
* Indication for emergency surgery

For rectal cancer patients:

* Contra-indication for MRI
* Absence of diagnostic pelvic MRI and/or contrast enhanced-CT thorax-abdomen
* Refusal of neoadjuvant treatment by the patient
* Absence of response assessment after (chemo)radiotherapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-07-13 (Actual); Primary Completion 2025-03 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Presence of lymph node metastases on FAPI PET/CT | <4 weeks from diagnosis for colon cancer and 10-17 weeks from diagnosis for rectal cancer
  Comparison: diagnostic contrast enhanced CT abdomen for colon cancer patients and diagnostic MRI for rectal cancer patients.
  Reference test: histopathology after surgery.
Number of positive regional lymph nodes (count) | <4 weeks from diagnosis for colon cancer and 10-17 weeks from diagnosis for rectal cancer
  Comparison: diagnostic contrast enhanced CT abdomen for colon cancer patients and diagnostic MRI for rectal cancer patients.
  Reference test: histopathology after surgery.
True malignant node (yes/no) | <4 weeks from diagnosis for colon cancer and 10-17 weeks from diagnosis for rectal cancer
  Comparison: diagnostic contrast enhanced CT abdomen for colon cancer patients and diagnostic MRI for rectal cancer patients Comparison: diagnostic contrast enhanced CT abdomen for colon cancer patients and MRI after neoadjuvant treatment for rectal cancer patients

SECONDARY OUTCOMES:
To describe additional findings on FAPI PET/CT i.e., structures with tracer uptake not including the primary tumour and/or regional lymph nodes. | <4 weeks from diagnosis
  Comparison: CT thorax-abdomen Reference test: none (biopsy of suspected lesions is not protocolized in this study) Parameters: presence of tracer uptake outside the area of primary tumour and lymph nodes (yes/no). If yes, description of the location, quantification of tracer uptake and descriptive comparison with standard diagnostic imaging.
To describe the correlation between tumour stroma in resected lymph node metastases and tracer uptake of lymph nodes on FAPI PET/CT. | <4 weeks from diagnosis for colon cancer and 10-17 weeks from diagnosis for rectal cancer
  Subgroup: patients who received resection of the tumour and lymph nodes. Parameters: visual and descriptive correlation between SUVmax and tumour stroma-related measures.
To describe the value of FAPI PET/CT on tumour response evaluation following neoadjuvant treatment. | 10-17 weeks from diagnosis for rectal cancer
  Subgroup: patients with rectal cancer Comparison: restaging MRI Reference test: histopathology after surgery Parameters: description and visualisation of delta SUV pre- and post-neoadjuvant therapy of the primary tumour and lymph nodes.

CONTACTS AND LOCATIONS:
Locations (2):
- Netherlands (2):
  - Noordwest ziekenhuisgroep, Alkmaar, North Holland
  - Netherlands Cancer Institute, Amsterdam, North Holland

IPD SHARING:
Plan to Share IPD: No